CLINICAL TRIAL: NCT05021133
Title: Tele-Navigation of Lung Cancer Screening
Brief Title: Tele-Navigation of Lung Cancer Screening (Tele-Navi LCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Wake Forest University Health Sciences (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mayuko Ito Fukunaga, Assistant Professor of Medicine, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H00022916; P50CA244693 (NIH)
Record Dates: First submitted 2021-08-10; First posted 2021-08-25 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
Keywords: lung cancer; cancer screening; health informatics
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-Navi LCS (Other): Tele-Navi of LCS includes: telehealth coaching from a Tele-Navigator for patients undergoing LCS
  Interventions: Behavioral: Tele-Navi LCS

INTERVENTIONS:
Behavioral: Tele-Navi LCS — Tele-Navi of LCS includes: telehealth coaching from a Tele-Navigator for patients undergoing LCS using a video or telephone call

SUMMARY:
Adherence to annual follow up is critical to achieving mortality benefits and optimizing cost-effectiveness of lung cancer screening (LCS). However, adherence to LCS follow-up in the real world is suboptimal. Using telehealth, the investigators will co-create Tele-Navigation of Lung Cancer Screening with patients and LCS stakeholders as an intervention to promote adherence of follow-up LCS. The investigators will then implement the Tele-Navi LCS intervention to a pilot sample of patients and evaluate its feasibility in the primary care setting. The investigators will measure the number of patient participants who completed Tele-Navi LCS and follow-up LCS within 180 days from Tele-Navi LCS.

ELIGIBILITY:
Inclusion Criteria:

* Is eligible for LDCT for LCS follow-up
* Has technology to complete study activities (e.g., video call visit)
* English speaker
* Has undergone LCS at UMMH
* Is overdue for LDCT follow-up

Exclusion Criteria:

* Has previous diagnosis of lung cancer
* Has active cancer diagnosis
* Is a nursing home or group care resident
* Is pregnant

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2025-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayuko Ito Fukunaga, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified (by HIPAA standards) dataset may be made available to the public with PI approval.
Supporting Information: Study Protocol

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 22 enrolled participants, 2 withdrew prior to the baseline survey.
Period: Overall Study
Arm/Group | Tele-Navi LCS
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Tele-Navi LCS: Tele-Navi of LCS includes telehealth coaching from a Tele-Navigator for patients undergoing LCS using a video or telephone call
Arm/Group | Tele-Navi LCS
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.5 [58.5 to 68.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Completion of Tele-Navi LCS
Description: Number of participants completed Tele-Navi LCS,
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-Navi LCS
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Completion of Follow-up LCS
Description: Number of participants who received a low-dose CT (LDCT) for LCS follow-up
Time Frame: 180 days
Population: 2 participants moved out from the healthcare system
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-Navi LCS
Number analyzed (Participants) | 18
Participants | 10

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed for each participant through study completion up to 180 days.
Description: No adverse event
Arm/Group | Tele-Navi LCS
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT05021133/Prot_SAP_000.pdf